CLINICAL TRIAL: NCT02797028
Title: Investigation of the Atherogenic Effects of Uric Acid-modified in Endothelial Dysfunction and the the Preventional Mechanism by Anthocyanidines
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yuan Zhang, Doctor of Medicine, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: No. 81402671
Record Dates: First submitted 2016-05-12; First posted 2016-06-13 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Cardiovascular Disease
Keywords: Hyperuricemia; endothelial function; anthocyanidins
MeSH Terms: conditions — Cardiovascular Diseases; Hyperuricemia | interventions — Anthocyanins; Allopurinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo capsule (Placebo Comparator): Simple hyperuricemia patients and with coronary heart disease in hospital. Double blind, randomized method. Control group taking placebo capsule
  Interventions: Dietary Supplement: Placebo capsule
- Anthocyanidins capsule (Experimental): Simple hyperuricemia patients and with coronary heart disease in hospital. Double blind, randomized method. The experimental group taking anthocyanins capsule.
  Interventions: Dietary Supplement: Anthocyanidins capsule
- Allopurinol (Experimental): The experimental group taking allopurinol.
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Dietary Supplement: Anthocyanidins capsule — Continuous intervention for 1 years, detect the indicators in the intervention of 0,6,12 months
  Arms: Anthocyanidins capsule
Dietary Supplement: Placebo capsule — Continuous intervention for 1 years, detect the indicators in the intervention of 0,6,12 months
  Arms: Placebo capsule
Drug: Allopurinol — Continuous intervention for 1 years, detect the indicators in the intervention of 0,6,12 months
  Arms: Allopurinol

SUMMARY:
The purpose of this study is to confirm the protective effect and mechanism of anthocyanins on hyperuricemia patients with Cardiovascular disease.

DETAILED DESCRIPTION:
Hyperuricemia patients who have the ability to complete the intervention study in the early stage of study were selected as the research subjects. A randomized controlled double blind control method was used to study the effect of one year of anthocyanins intervention. Serum UA levels, oxidative stress, AGEs, and endothelial function are detecting in patients with hyperuricemia who were treated with anthocyanins and placebo. Providing scientific basis of anthocyanins for the treatment with hyperuricemia and delaying atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Serum uric acid >420μmol/L (7mg/dL) in male, >360μmol/L (6mg/dL) in female identified as hyperuricemia patients.

Exclusion Criteria:

* Age more than 60 years and less than 30 years old;
* acute infection, tumor, recent surgery, need for hemodialysis and autoimmune diseases.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of serum uric acid levels in all patients | up to 1 months
  Serum uric acid (mg/dl) is determined by Uric Acid kit on an automated system.

SECONDARY OUTCOMES:
Measurement of advanced glycation end products and its receptor level in all patients | up to 2 months
  Advanced glycation end products and its receptor level are determined by high efficiency liquid chromatography.

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Guangzhou Military Command of People's Liberation Army, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Davignon J, Ganz P. Role of endothelial dysfunction in atherosclerosis. Circulation. 2004 Jun 15;109(23 Suppl 1):III27-32. doi: 10.1161/01.CIR.0000131515.03336.f8. PMID 15198963
- [Background] Gimbrone MA Jr. Endothelial dysfunction and atherosclerosis. J Card Surg. 1989 Jun;4(2):180-3. doi: 10.1111/j.1540-8191.1989.tb00275.x. PMID 2519996
- [Background] Verma S, Anderson TJ. Fundamentals of endothelial function for the clinical cardiologist. Circulation. 2002 Feb 5;105(5):546-9. doi: 10.1161/hc0502.104540. No abstract available. PMID 11827916
- [Background] D'Marco L, Garcia I, Vega C. [Uric acid, atherosclerosis and vascular calcifications in chronic kidney disease]. Invest Clin. 2012 Mar;53(1):52-9. Spanish. PMID 22524108
- [Background] Feig DI, Kang DH, Johnson RJ. Uric acid and cardiovascular risk. N Engl J Med. 2008 Oct 23;359(17):1811-21. doi: 10.1056/NEJMra0800885. No abstract available. PMID 18946066
- [Background] Li C, Han L, Levin AM, Song H, Yan S, Wang Y, Wang Y, Meng D, Lv S, Ji Y, Xu X, Liu X, Wang Y, Zhou L, Miao Z, Mi QS. Multiple single nucleotide polymorphisms in the human urate transporter 1 (hURAT1) gene are associated with hyperuricaemia in Han Chinese. J Med Genet. 2010 Mar;47(3):204-10. doi: 10.1136/jmg.2009.068619. Epub 2009 Oct 14. PMID 19833602